CLINICAL TRIAL: NCT06449976
Title: Application and Clinical Evaluation of Longitudinal Chromatic Aberration Technique in Ophthalmology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: BeijingTH-202405
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-05

CONDITIONS: Longitudinal Chromatic Aberration; Blue Light Defocus Manipulation
Keywords: Longitudinal chromatic aberration; Reading efficiency; Visual function; Visual fatigue; Fundus blood flow; Axial length; Total refraction difference value
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Intervention Model Description: This study is designed with a total of four groups, where participants will sequentially and randomly undergo all the intervention procedures.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Blue Light 0D Defocus Group (Experimental): This is the group that performs visual evoked tasks using videos and texts that are not defocused in the blue channel. In this group, the impact of standard video modes on the axial length of the eye, refractive fatigue, and visual function is assessed, including but not limited to indicators such as reading efficiency, blinking detection, and retinal fundus blood flow.
  Interventions: Behavioral: blue light defocus and blue light filtering
- Blue Light 1D Defocus Group (Experimental): Group using blue channel defocused 1D videos and texts for visual evoked tasks. Participants will engage in a 50-minute visual evoked task using videos and texts processed with 1D blue channel. The impact of standard video mode on axial length of the eye, refractive labor, and visual function will be assessed, including but not limited to indicators such as reading efficiency, blinking detection, and retinal fundus blood flow.
  Interventions: Behavioral: blue light defocus and blue light filtering
- Blue Light 2D Defocus Group (Experimental): The group uses blue channel defocused 2D videos and texts for visual evoked tasks. Participants will undergo a 50-minute visual evoked task using videos and texts processed with the 2D blue channel. The effects of standard video mode on the eye's axial length, refractive labor, and visual function are assessed, including but not limited to indicators such as reading efficiency, blinking detection, and retinal fundus blood flow.
  Interventions: Behavioral: blue light defocus and blue light filtering
- Blue Light 1D Defocus with Partial Filtration Group (Experimental): The group uses videos and texts processed with the blue channel 1D defocus and 30% blue light filtering for visual evoked tasks. Participants will engage in a 50-minute visual evoked task using videos and texts that have been processed with the 1D blue channel and partially filtered for blue light. The impact of the standard video mode on the eye's axial length, refractive labor, and visual function is evaluated, including but not limited to indicators such as reading efficiency, blinking detection, and retinal fundus blood flow.
  Interventions: Behavioral: blue light defocus and blue light filtering

INTERVENTIONS:
Behavioral: blue light defocus and blue light filtering — Subjects are asked to watch a terminal display device for 50 minutes, featuring texts and videos with different defocusing treatments. Specifically, they will start by watching text for 5 minutes, followed by 40 minutes of video, and then another 5 minutes of text, totaling a visual task duration of 50 minutes. The participants will complete a total of 4 sets of tests in a random order.

SUMMARY:
Our study aims to delve into the effects of shifting the focal point of blue light from video or text displayed on a terminal screen forward on the axial length of the eye, ocular blood flow, visual fatigue, and visual function, that is, its relationship with Video Display Terminal (VDT) syndrome and myopia. By examining the decoding ability of the adult subjects' retina to the clarity of the signal, we will attempt to develop a novel, non-invasive strategy to curb the elongation of the eyeball associated with myopia. Concurrently, we will also focus on the pathophysiological mechanisms underlying VDT syndrome and explore its potential link to the progression of myopia, providing new scientific evidence for the prevention and treatment of this ocular condition. This research is expected to provide robust support for addressing the global issue of myopia and the health challenges posed by VDT syndrome. Ultimately, by integrating global eye health issues with the challenges brought about by VDT syndrome, we will propose intervention and prevention strategies, offering new insights for the advancement of ophthalmology and public health sectors, thereby promoting visual acuity and ocular health for the population.

ELIGIBILITY:
Inclusion Criteria:

1. Adult population, regardless of gender
2. Refractive error is less than or equal to -2.5D and both eyes achieve corrected visual acuity of 0.8 or higher.
3. Normal intraocular pressure with no organic pathology.
4. No apparent symptoms of dry eye.
5. Willing to cooperate to complete all the tests.
6. Voluntarily signing the informed consent form.

Exclusion Criteria:

1. Individuals with strabismus and amblyopia exist.
2. Suffering from congenital eye conditions such as congenital cataracts or congenital retinal diseases.
3. Those who have undergone intraocular surgery (such as cataract removal, intraocular lens implantation, etc.).
4. Individuals with refractive media opacity (such as corneal lesions, lens opacity, etc.).
5. Abnormal intraocular pressure (IOP) (IOP < 10 mmHg or IOP > 21 mmHg, or a bilateral IOP difference of ≥5 mmHg).
6. Only one eye meets the inclusion criteria.
7. Active corneal infections such as bacterial, fungal, viral, or other acute or chronic anterior segment inflammations.
8. Currently using medications that may lead to dry eye or affect vision and corneal curvature.
9. Other ocular conditions, such as dacryocystitis, eyelid disorders and abnormalities, abnormal intraocular pressure, and glaucoma.
10. Unable to undergo regular eye examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Ocular Fundus Blood Flow | The total duration of the visual task is 50 minutes. Retinal blood flow is measured for each subject at 0 minutes, 25 minutes, and 50 minutes during the visual task, resulting in a
  The study measured the sub foveal choroidal thickness, superficial vessel complex (SVC) density, and deep vessel complex (DVC) density, analyzing changes in retinal blood flow under the two modes.

SECONDARY OUTCOMES:
Visual fatigue | Each participant will complete the visual fatigue questionnaire, followed immediately by a VEP task, and then re-assess visual fatigue immediately afterward. This sequence will occur twice per group, totaling eight assessments per participant.
  The visual fatigue questionnaire utilized in this study consists of a self-report survey with a total of 19 items. It is designed to comprehensively assess the severity of visual fatigue symptoms, with a scoring system ranging from 1 to 7. Higher scores indicate more severe symptoms, encompassing three primary domains: ocular symptoms, visual discomfort, and psychological aspects triggered by visual fatigue.
Measurement of Accommodative Sensitivity with Flip-Chart Post-VEP Tasks | Each participant will have five measurements: a baseline, and four post-VEP tasks, with immediate flipchart tests after each task.
  This clinical study involves the assessment of accommodative sensitivity for both monocular and binocular vision using a flip-chart immediately following each visual evoked potential (VEP) task. The measurement will quantify the number of optotypes correctly identified within one minute, indicative of the subject's accommodative capacity.
Blink Frequency | Blink frequency 3 minutes after the start of each visual evoked task and 3 minutes before the end.
  Use electronic devices to record the number of clicks within 3 minutes and calculate the frequency.
Reading efficiency | The test was recorded 5 minutes after the start and 10 minutes before the end.
  The number pairs were read in the first and last 5 minutes of the visual evoked task, and the number of number pairs read per minute was counted.
AC/A Ratio Measurement Post-VEP Tasks | Each participant will undergo five AC/A ratio measurements: at baseline and immediately after each of four VEP tasks.
  This study involves the measurement of the AC/A ratio, which is a critical parameter in binocular vision assessment, reflecting the relationship between accommodation (focus adjustment) and convergence (ocular alignment). The AC/A ratio will be determined using the prism bar technique, which involve adding lenses to stimulate accommodation and measuring the resulting changes in convergence.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospitol, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No